CLINICAL TRIAL: NCT01016860
Title: A Phase I/IB Study of OSI-906 and Irinotecan in Patients With Advanced Cancer With Expanded Cohorts of Patients With Colorectal Cancer Stratified by the OSI-906 Integrated Classifier
Brief Title: OSI-906 and Irinotecan in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was discontinued due to a shown lack of efficacy in the investigational agent
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0705.cc; NCI-2011-03204 (Other: National Cancer Institute)
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer
Keywords: OSI-906, irinotecan, colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OSI-906 and/or irinotecan (Experimental): Dose Escalation Phase: Treatment for Cycle 1 will commence on Day -3 of a 21-day cycle (3 weeks) when a single dose OSI-906 is given with full pharmacokinetics(PK) sampling at predetermined time points. Irinotecan will be administered intravenously over 90 minutes on Day 1 and Day 8 with full PK sampling on Day 1. The institution of oral dosing of OSI-906 2-4, 8-10, 15-17 (for cycle 1 only) will be given followed by full PK sampling of both drugs on Day 8. Pre-dose samples of OSI-906 will be drawn on Cycle 1 Days 8, 10, 15, 17 and Cycle 2 Days 1, 8, 10, 15 and 17. For Cycle 2 and thereafter, both drugs will be administered starting on Day 1.
  Interventions: Drug: OSI-906; Drug: irinotecan

INTERVENTIONS:
Drug: OSI-906 — OSI-906 will be given orally in tablets for one dose starting on Cycle 1 Day-3 then on Cycle 1 Day 2-4, 8-10 and 15-17. Cycle is 21 days. Subsequent cycles, dosing will start be Day 1-3, 8-10 and 15-17
  Other Names: Linsitinib
Drug: irinotecan — Irinotecan will be administered IV over 90 minutes on Day 1 and 8 of a 21-day cycle
  Other Names: Camptosar

SUMMARY:
This study plans to learn more about an investigational drug called OSI-906. OSI-906 is being looked at to see if it could be a treatment for advanced cancer. "The FDA is the U.S. government agency that reviews the results of research of drugs and decides if it can be sold in the U.S. OSI-906 has been given to over 185 people with cancer.

DETAILED DESCRIPTION:
This study plans to learn more about an investigational drug called OSI-906. OSI-906 is being looked at to see if it could be a treatment for advanced cancer.

Subjects will also receive a drug called irinotecan (also called Camptosar®). This drug is FDA approved for the treatment of metastatic colon cancer and some other types of cancer. The study drug and irinotecan have never been tested together in humans. It is unknown if the combination will be safe and/or effective in the treatment of human cancers.

The purpose of this study is to find the answers to the following research questions:

* What is the highest dose of the study drug that can be given to subjects in combination with irinotecan without causing side effects that are too severe?
* How is the combination of the study drug and irinotecan handled in the blood of subjects with advanced cancer? Does either the study drug or irinotecan have an effect on how the other works?
* What are the most common side effects of the study drug and irinotecan when given together to subjects with advanced cancer?
* Is the combination of the study drug and irinotecan effective in stopping the growth or shrinking the size of your tumor?

ELIGIBILITY:
Inclusion Criteria:

• Dose Escalation Phase: Histological or cytopathological diagnosis of an advanced cancer that is refractory to standard therapy or for which no standard therapy exists.

Irinotecan must be listed in the Compendia for reimbursement, ie. colorectal cancer; lung cancer; gastric; esophageal, cervical and ovarian cancer.

* Cohort Expansion Phase: Histological or cytopathological diagnosis of advanced colorectal cancer with known Kirsten rat sarcoma (KRAS) mutation status. All patients must have received and progressed or be intolerable of first-line therapy with an oxaliplatin-containing regimen. Patients must be screened using the OSI-906 integrated classifier.
* Cohort 1 (12 patients): Window of opportunity cohort: Patients with a score of at least 4 out of 5 by the OSI-906 integrated classifier who are irinotecan-naive will receive OSI-906 as a single agent until disease progression. Patients must be non surgically resectable or not a surgical candidate because of comorbid conditions. At disease progression, if the patient had a best response of at least stable disease for 3 cycles (9 weeks), irinotecan may be added to OSI-906.
* Cohort 2: (16 patients: 8 KRAS wild-type (WT) and 8 KRAS Mutant(MT). Patients who have score of less than 4 by the OSI-906 integrated classifier will have OSI-906 added to irinotecan on disease progression to irinotecan (patients that are KRAS WT will have received cetuximab with irinotecan). Patients who are treated in the dose escalation phase at the recommended phase II dose of the combination and meet the criteria for Cohort 2 of the expanded phase may be counted towards the dose expansion patient numbers.
* Age ≥18 years old
* Patients must have an Eastern Co-operative oncology group (ECOG) performance status of 0-1
* Life expectancy of at least three months.
* Adequate hematological function and bone marrow reserve:

Hematopoetic: Neutrophil count ≥ 1.5 x 109/L (1,500/mm3), Platelet count ≥ 75 x 109/L, Hemoglobin ≥ 9.0g/dL

* Adequate hepatic and renal function Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 fold upper limit of normal (ULN) Bilirubin ≤ 1.5 X ULN Creatinine ≤ 1.5 fold ULN or calculated creatinine clearance, using the Cockcroft-Gault formula > 60 mL/min, if just below 60 mL/min then Glomerular Filtration Rate > 60 mL/min as determined by 24 hour urine collection
* Measurable (according to Response Evaluation Criteria in Solid Tumors (RECIST) Criteria in the dose expansion cohorts or measurable /evaluable disease in the Dose Escalation phase,
* Ability to understand the requirements of the study, provide written informed consent and comply with the study protocol procedures.

A: Documentation of KRAS status must be performed prior to enrollment.

Exclusion Criteria:

* Concurrent symptomatic central nervous system involvement, brain or meningeal metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, uncontrolled diabetes, uncontrollable hypertension or psychiatric illness/social situations that would limit compliance with study requirements
* Documented history of diabetes
* Corrected QT (QTc) interval > 450 msec at baseline
* Drugs with a Risk of Causing corrected QT interval Prolongation: Drugs that have a risk of causing QT interval prolongation are prohibited within 14 days prior to Day 1 dosing and while on study to avoid exacerbation of any OSI-906 potential side effects
* Known positive serology for the human immunodeficiency virus (HIV), Hepatitis B and/or Hepatitis C
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Gastrointestinal tract disease (including peptic ulcer disease) or prior surgery resulting in an inability to take oral medications
* Patients may have had prior therapy, providing the following conditions are met:

Chemotherapy: A minimum of 3 weeks (4 weeks for carboplatin or investigational anticancer agents and 6 weeks for nitrosoureas and mitomycin C) must have elapsed between the end of treatment and start of treatment. Patients must have recovered from any treatment-related toxicities (except for alopecia, fatigue, and grade 1 neurotoxicity) prior to start of treatment.

Hormonal therapy: Patients may have had prior anticancer hormonal therapy provided it is discontinued prior to start of treatment. However, patients with prostate cancer with evidence of progressive disease may continue on therapy that produces medical castration (eg, goserelin or leuprorelin), provided this therapy was commenced at least 3 months earlier.

Radiation: Patients may have had prior radiation therapy provided they have recovered from the acute, toxic effects of radiotherapy prior to start of treatment. A minimum of 21 days must have elapsed between the end of radiotherapy and start of treatment if the radiation affected more than 25% of bone marrow otherwise a 14 days wash out is required.

Surgery: Previous surgery is permitted provided that wound healing has occurred prior to start of treatment.

• Laboratory results: international normalized ratio (INR) ≥ 1.5 X ULN and activated partial thromboplastin time (aPTT) ≥ 1.5 X ULN

Fasting blood glucose of >125mg/dL at baseline and on Day 1 of dosing.

* Women who are pregnant or breast feeding because of teratogenic potential.
* Women of childbearing potential in whom pregnancy cannot be excluded or who are not using an adequate method of contraception because of teratogenic potential.
* Prior documented hypersensitivity to irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and the recommend phase II dose (RP2D) for the combination of irinotecan and OSI-906 in patients with advanced cancer. | Up to 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Leong, M.D, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Davis SL, Eckhardt SG, Diamond JR, Messersmith WA, Dasari A, Weekes CD, Lieu CH, Kane M, Choon Tan A, Pitts TM, Leong S. A Phase I Dose-Escalation Study of Linsitinib (OSI-906), a Small-Molecule Dual Insulin-Like Growth Factor-1 Receptor/Insulin Receptor Kinase Inhibitor, in Combination with Irinotecan in Patients with Advanced Cancer. Oncologist. 2018 Dec;23(12):1409-e140. doi: 10.1634/theoncologist.2018-0315. Epub 2018 Aug 23. PMID 30139840